CLINICAL TRIAL: NCT06125327
Title: A Randomized, Double-blind, Placebo-controlled Phase II/III Trial Evaluating the Efficacy and Safety of Sufenidone (SC1011) Tablets in Patients With Idiopathic Pulmonary Fibrosis (IPF).
Brief Title: SC1011 Twice Daily vs Placebo in Patients Diagnosed With Idiopathic Pulmonary Fibrosis (IPF)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Guangzhou JOYO Pharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JYP1011M201
Record Dates: First submitted 2023-11-04; First posted 2023-11-09 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis; Lung Diseases; Respiratory Tract Diseases
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Lung Diseases; Respiratory Tract Diseases | interventions — Bulk Drugs

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Comparator (Placebo Comparator): Idiopathic pulmonary fibrosis (IPF) patients were administered placebo matching SC1011 taken orally as tablets (matching the respective SC1011 tablets) twice daily, in the morning and in the evening for 52 weeks.
  Interventions: Drug: Placebo comparator
- SC1011 200mg (Experimental): Idiopathic pulmonary fibrosis (IPF) patients were administered SC1011 taken orally as tablets twice daily(200mg daily), in the morning and in the evening for 52 weeks.
  Interventions: Drug: SC1011

INTERVENTIONS:
Drug: SC1011 — Patients receive the dose of SC1011 tablets orally twice daily (b.i.d) for 52 weeks.
  Other Names: Active Drug
  Arms: SC1011 200mg
Drug: Placebo comparator — Patients receive the dose of placebo orally twice daily (b.i.d) for 52 weeks.
  Other Names: comparator
  Arms: Placebo Comparator

SUMMARY:
Evaluating Sufenidone (SC1011) in IPF patients for efficacy and safety. Includes screening, treatment, and follow-up, with FVC decline and health checks.

DETAILED DESCRIPTION:
Randomized, double-blind study comparing Sufenidone (SC1011) and placebo in IPF patients, with interim analysis at 26 weeks to select the optimal dose for a 52-week treatment period followed by 4-week safety monitoring

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and sign written informed consent.
* The diagnosis time of IPF before enrollment was less than 5 years.
* Combination of High Resolution Computerized Tomography (HRCT) pattern, and if available surgical lung biopsy pattern, as assessed by central reviewers, are consistent with diagnosis of IPF.
* Dlco (corrected for Hb): 30%-90% predicted of normal.
* FVC>= 50% predicted of normal.

Exclusion Criteria:

* Forced expiratory volume in one second (FEV1)/FVC ratio <0.7 after administration of bronchodilator at Screening
* Expected to receive a lung transplant within 1 year from randomization or, for patients at sites in the United States, on a lung transplant waiting list at randomization.
* Known explanation for interstitial lung disease
* History of asthma or chronic obstructive pulmonary disease
* Active infection
* Ongoing IPF treatments including investigational therapy, immunosuppressants, and cytokine modulating agents
* History of unstable or deteriorating cardiac or pulmonary disease (other than IPF) within the previous 6 months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Annual Rate of Decline in Forced Vital Capacity (FVC) Over 52 Weeks | Primary Outcome measures will be assessed at baseline and again at 52 weeks.
  Forced vital capacity (FVC) is the total amount of air exhaled during the lung function test. For this endpoint reported means represent the adjusted rate.

SECONDARY OUTCOMES:
Change From Baseline in Saint-George's Respiratory Questionnaire (SGRQ) Total Score at 52 Weeks | Baseline and 52 weeks
  SGRQ is a health-related quality of life questionnaire divided into 3 components : symptoms, activity and impact.The total score (summed weights) can range from 0 to 100 with a lower score denoting a better health status. Means provided are the adjusted means based on all analyzed patients in the model (not only patients with a baseline and measurement at week 52)
Time to First Acute Idiopathic Pulmonary Fibrosis (IPF) Exacerbation. | Secondary outcome measures will be assessed at baseline and again at 52 weeks.
  Due to rare events, the median of time to event is not calculable, thus the percentages of patients with (IPF) exacerbation are reported and represented as a key secondary endpoint.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No